CLINICAL TRIAL: NCT06642194
Title: The Effectiveness of Sunnah on Sleeping on Sleep Quality, Fatigue, Depression and
Brief Title: The Effectiveness of Sunnah on Sleeping on Sleep Quality, Fatigue, Depression and Anxiety Among Patient Undegroing Hemodialysis
Acronym: sleeping
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Muhammadiyah Yogyakarta (Other)
Responsible Party: Principal Investigator, Erna Rochmawati, Professor, Universitas Muhammadiyah Yogyakarta
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Sunnah on sleeping
Record Dates: First submitted 2024-10-13; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Sleep Quality; Fatigue; Anxiety; Depression
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Fatigue; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education on sunnah of sleeping (Experimental): Participants in the experimental group received education on sunnah of sleeping for two weeks. The interventions had three session which conducted between 40-60 minutes per session. The session include: 1) introducing the research objectives, definition and benefits on sunnah of sleeping; 2) steps in sunnah of sleeping 3) providing mp3 and prayers beads to facilitate Qur'an recitation and zikr. These surat was chosen because the portion of surat concentrate on the absolute divinity of Allah and Allah's blessings to His creatures. The steps in sunnah of sleeping can be performed approximately about 10-15 minutes about 30 minutes prior to sleep.
  Interventions: Behavioral: Education on sunnah of sleeping
- Control group (No Intervention): While the experiment group received education on sunnah of sleeping, the control group received standard care without receiving the education on sunnah of sleeping.

INTERVENTIONS:
Behavioral: Education on sunnah of sleeping — The interventions had three session which conducted between 40-60 minutes per session. The session include: 1) introducing the research objectives, definition and benefits on sunnah of sleeping; 2) steps in sunnah of sleeping (early bedtime and early wake up time; perform ablution (wudoo) before going to bed and supplicate; dusting and cleaning the bed before sleeping; sleep position; turning off light before sleep; cover mouth when yawning and reciting some verses such as Ayat Kursi, Al-Ikhlas, Al-Falq and An-Nas); 3) providing mp3 and prayers beads to facilitate Qur'an recitation and zikr. These surat was chosen because the portion of surat concentrate on the absolute divinity of Allah and Allah's blessings to His creatures. The surat brings every Muslim the closeness to Allah, the calmness of the soul, and the cure for many physical and psychological diseases. The steps in sunnah of sleeping can be performed approximately about 10-15 minutes about 30 minutes prior to sleep.
  Arms: Education on sunnah of sleeping

SUMMARY:
This study to examine the effects of implementation sunnah on sleeping on sleep quality, sleep time receiving a slow stroke back massage on fatigue and quality of life among participants undergoing maintenance hemodialysis will be applied. The study will be conducted at the hemodialysis unit of a medical center in a central part of Indonesia. To determine the sample size at a 95% confidence level and 80% test power, with a mean difference of at least 0.72 and a standard deviation of 1.22 in the intervention group and 1.22 in the control group, based on the study of [17] and according to the sample size formula, we determined a requirement of 205participants in each group. Forty participants were recruited and allocated to either the experimental group (n=25) or the control group (n = 25).

Participants will be recruited if they were: (i) 18 years of age or over; (ii) under- going hemodialysis for a minimum of three months; (iii) undergoing maintenance hemodialysis; (iv) diagnosed with a maximum of two comorbidities; (v) affiliated to Islam; and (vi) not hearing-impaired. Participants were excluded if they had, (i) muscle problems, and (3) unstable vital signs. A thorough review of participant charts will be performed to confirm they met the inclusion and exclusion criteria. Participants then will be randomly assigned to two different groups based on their hemodialysis schedule.

The measurement of demographic and illness-related characteristics; the Functional Assessment of Chronic Illness Therapy-fatigue (FACIT-fatigue) and Pitssburg Sleep Quality Index (PSQI) will be conducted at the baseline and after the fourth week. The FACIT-fatigue scale was used to measure participant fatigue. FACIT-fatigue has 13 items to assess fatigue and its impact on functioning and daily activities in a number of chronic diseases, with five-point response options from 0 to 4. The total score ranges from 0 to 52, where a higher total score reflects less fatigue. The items include tiredness, listlessness, weakness, lack of energy, and impact on daily. In the study, we will use a validated Indonesian version of FACIT-fatigue. This version has been tested on 52 participants by Sihombing et al 2016 with CKD and has good internal reliability with a Cronbach's alpha of 0.62 (20). The PSQI has been translated and tested for validity and reliability by Setyowati & Chung (2021). The Cronbach alpha for Indonesian version of PSQI is 0.72 which means that the Indonesian version of PSQI has adequate reliability (21).

ELIGIBILITY:
Inclusion Criteria:

Participants undergoing hemodialysis were recruited if they were: (1) 18 years of age or over; (2) undergoing maintenance hemodialysis twice a week for a minimum of three months; (3) affiliated to Islam, and (4) not hearing-impaired

Exclusion Criteria:

* Participants were excluded if they had unstable vital signs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Sleep quality | Will be measured at base line and after three weeks, prior to hemodialysis procedure
  The Pittsburgh Sleep Quality Index (PSQI) has 19 items to assess sleep quality which can be categorized to seven domain; (1) sleep quality; (2) sleep latency; (3) sleep duration; (4) habitual sleep efficiency; (5) sleep disturbance; (6) sleep medication and (7) daytime sleep disturbance. The total score 1-21, where a higher total score reflect lower sleep quality.
Fatigue | Will be measured at base line and after three weeks, prior to hemodialysis procedure
  The FSS was used to assess participant's fatigue and its impact to activities and life style. The FSS has nine items, with response options from 1-7, where a higher total score reflects higher fatigue

CONTACTS AND LOCATIONS:
Locations (1):
- RS PKU Muhammadiyah Yogyakarta, Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided
The study will be shared upon request